CLINICAL TRIAL: NCT05601011
Title: Changes of Clinical Characteristics and Tear Film Biomarkers Following FS-LASIK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RS
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — basal tears
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to analyze the clinical and tear molecular profile up to 6 months after FS-LASIK surgery

DETAILED DESCRIPTION:
FS-LASIK is a refractive surgery technique widely used in China. To explore the role of inflammation and nerve in the occurrence and development of dry eyes after FS-LASIK by dynamically observing the ocular surface characteristics and the levels of inflammatory factors and neurotransmitters in the early and late stage after FS-LASIK.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who preparing for FS-LASIK with age between 18 and 45 years old
2. Any gender
3. Provision of written informed consent.

Exclusion Criteria:

1. active ocular infection, ocular inflammation, active ocular allergy, severe blepharitis or obvious inflammation of the eyelid margin.
2. Pregnant and lactating women, or those planning a pregnancy over the course of the study
3. Uncontrolled systemic disease
4. Suffer from diseases that may affect corneal nerves, such as keratoconus, trigeminal neuralgia, allergic conjunctivitis, etc.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: All patients from Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-10-19 (Estimated); Study Completion 2023-10-19 (Estimated)

PRIMARY OUTCOMES:
ocular surface disease index (OSDI) | from Pre-surgery to 6 months after surgery
  OSDI is one of the most frequently used questionnaires for evaluation of dry eye disease (DED). This includes 12 questions which measure the frequency of symptoms over the recent week, and the scores range from 0 to 100.
Tear break-up time (TBUT)(s) | from Pre-surgery to 6 months after surgery
  BUT is the time from normal blinking to the first appearance of a break in the tear film.
Corneal fluorescein staining (CFS) | from Pre-surgery to 6 months after surgery
  The degree of fluorescein staining of the cornea was evaluated using the National Eye Institute (NEI) scale of five corneal regions (central, superior, temporal, nasal, and inferior). The scores range from 0 to 15.
Schirmer Ⅰ test (SⅠt) (mm/5 minutes) | from Pre-surgery to 6 months after surgery
  The Schirmer I test is performed using sterile strips without anesthesia. The strips are placed in the lateral part of the inferior fornix of the eye for 5min and the extent of tear flow down was measured in millimeters.

SECONDARY OUTCOMES:
the concentration of Interleukin-1β（IL-1β) (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-1β levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-6 (IL-6) (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-6 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-10 (IL-10) (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-10 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-23 (IL-23) (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-23 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-17A (IL-17A) (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-17A levels will be quantified by Luminex immunoassay.
the concentration of tumor necrosis factor-α (TNF-α)(pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. TNF-α levels will be quantified by Luminex immunoassay.
the concentration of interferon-γ (IFN-γ)(pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IFN-γ levels will be quantified by Luminex immunoassay
the concentration of granulocyte-macrophage colony-stimulating factor (GM-CSF)(pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. GM-CSF levels will be quantified by Luminex immunoassay.
the concentration of substance P (SP)(pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. SP levels will be quantified by Luminex immunoassay.
the concentration of alpha-melanocyte-stimulating hormone (α-MSH) (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. α-MSH levels will be quantified by Luminex immunoassay.
the concentration of β-endorphin (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. β-endorphin levels will be quantified by Luminex immunoassay.
the concentration of neurotensin (pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. β-endorphin levels will be quantified by Luminex immunoassay.
the concentration of oxytocin(pg/ml) | from Pre-surgery to 6 months after surgery
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. oxytocin levels will be quantified by Luminex immunoassay.
Lissamine green staining | from Pre-surgery to 6 months after surgery
  To grade the temporal zone, the subject looks nasally; to grade the nasal zone the subject looks temporally. The upper and lower conjunctiva can also be graded.
meibomian gland dropout rate | from Pre-surgery to 6 months after surgery
  grade 0: no gland atrophy; grade 1: ≤1/3 gland atrophy; grade 2: 1/3 to 2/3 gland atrophy；grade 3: >2/3 gland atrophy.
corneal sensitivity (range, 60-0 mm) | from Pre-surgery to 6 months after surgery
  Corneal sensitivity will be measured in the right eye only using the Cochet-Bonnet aesthesiometer and the ascending method of limits to determine the threshold of stimulus detection.
sub-basal corneal nerve density (mm/mm2) | from Pre-surgery to 6 months after surgery
  Sub-basal corneal nerve plexus image will be acquired using a laser scanning confocal microscope.
numerical rating scale (NRS) | from Pre-surgery to 6 months after surgery
  The NRS was used to evaluate ocular pain and consists of a numbered line from 0 to 10 scores that measures pain intensity: 0-1: no pain; 2-4: mild pain; 5-7: moderate pain; and 8-10: severe pain.
NPSI-Eye (range 0-100 score) | from Pre-surgery to 6 months after surgery
  Neuropathic Pain Symptom Inventory modified for the Eye (NPSI-Eye) (range 0-100 over a 24-hour recall period)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No